CLINICAL TRIAL: NCT05796167
Title: Does Pimavanserin (Nuplazid) Improve Sleep in Patients With Parkinson Disease Psychosis? A Pilot Study
Brief Title: Pimavanserin for Sleep in Parkinson Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The PI did not have eligible candidates. Therefore, Acadia Pharmaceuticals (the sponsor) closed the study.
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-02-723-205; 1396075255 (Other: Acadia Pharmaceuticals Inc)
Record Dates: First submitted 2023-01-31; First posted 2023-04-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: sleep; visual hallucinations; delusions
MeSH Terms: conditions — Parkinson Disease; Hallucinations; Delusions | interventions — pimavanserin

STUDY DESIGN:
Intervention Model Description: self-control, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pimavanserin (Nuplazid) (Experimental): Pimavanserin (Nuplazid) 34 mg oral capsules once a day for 6 weeks for patients with Parkinson disease psychosis (e.g., visual hallucinations, delusions) and sleep problems
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin (Nuplazid) 34 mg oral capsules once a day for 6 weeks
  Other Names: Nuplazid

SUMMARY:
This pilot, self-control study is for patients with Parkinson's Disease (PD) psychosis (e.g., visual hallucinations, delusions) and sleep problems.

DETAILED DESCRIPTION:
This is a feasibility study to determine whether pimavanserin improves sleep quality in patients with PD and visual hallucinations/delusions.

Patients will complete a Screening Visit to assess eligibility to participate in the study.

For more information, please contact Sofya Glazman, a study coordinator, at sofya.glazman@downstate.edu

ELIGIBILITY:
Inclusion criteria:

1. Has a diagnosis of idiopathic PD according to UK (United Kingdom) PD Society Brain Bank diagnostic criteria
2. Has a history of hallucinations or delusions associated with PD
3. Has a history of sleep disturbance
4. Is between the ages of 40 and 85
5. Has been on a stable dose of all PD medications for at least 30 days prior to enrolment

Exclusion criteria

1. Has evidence of an atypical or secondary parkinsonian disorder
2. Has a contraindication to taking pimavanserin
3. Has contraindication to PSG
4. There has been a change to patient's neuropsychiatric medications including dopaminergic medications (Sinemet, dopamine agonists, MAO(monoamine oxidaze)-B inhibitors), SSRIs (Selective Serotonin Reuptake Inhibitors), SNRIs (Serotonin and Norepinephrine Reuptake Inhibitors), dopamine-blocking agents, anti-epileptics, anticholinergics, or benzodiazepines for at least 30 days prior to enrollment
5. Has traveled through 3 or more time zones within 60 days prior to study screening
6. Patient is a night-shift worker

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Effect of pimavanserin on sleep fragmentation | 6 weeks
  Number of arousals and the arousal index (arousals per hour of sleep) measured on polysomnography

SECONDARY OUTCOMES:
Effect of pimavanserin on REM (Rapid Eye Movements) sleep behavior disorder | 6 weeks
  Presence fo REM sleep without atonia (RWA) on polysomnograophy
Effect of pimavanserin on sleep latency | 6 weeks
  Time to first epoch on polysomnography
Effect of pimavanserin on total sleep time | 6 weeks
  Total sleep time measured on polysomnography
Effect of pimavanserin on sleep efficiency | 6 weeks
  Sleep Efficiency Index in percent is the ratio of total sleep time (based on polysomnography recordings) to time in bed
Effect of pimavanserin on time in each sleep stage | 6 weeks
  Time in each sleep stage as measured on polysomnography
Effect of pimavanserin on subjective measure of REM Sleep behavior disorder | 6 weeks
  RBDSQ (REM (Rapid Eye Movements) Sleep Behavior Disorder Screening Questionnaire to assess the most prominent clinical features of RBD. It is a 10-item, patient self-rating instrument with short questions to be answered by either 'yes' or 'no'.
Effect of pimavanserin on subjective measures of sleep | 6 weeks
  PDSS-2 (Parkinson's Disease Sleep Scale Version 2) total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance). Scores > 18 are considered as relevant sleep disturbances
Effect of pimavanserin on subjective measures of fatigue | 6 weeks
  PFS-16 (Parkinson's disease Fatigue Scale): 16-item scale with the following scoring for each item: strong disagree -1, disagree - 2, neither agree or disagree - 3, agree - 4, strongly agree - 5; with overall score of ≥8 indicates the presence of significant fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Christian J Amlang, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Health Sciences University, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT05796167/Prot_001.pdf